CLINICAL TRIAL: NCT04224766
Title: Comparison Between Interscalene and Combined Costoclavicular-suprascapular Blocks for Arthroscopic Shoulder Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, mohamed talaat mohamed mohamed, assistant lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 17200124
Record Dates: First submitted 2020-01-06; First posted 2020-01-13 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Shoulder Surgery; Regional Anesthesia Morbidity
Keywords: regional anesthesia; interscalene brachial plexus block; suprascapular and costoclavicular blocks

STUDY DESIGN:
Intervention Model Description: 2 groups of patients. Randomization into groups SSNP + costoclavicular or ISBPB as per randomization list, for a total of 50 patients.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- suprascapular nerve block with costoclavicular infraclavicular (Experimental): Single shot US-guided suprascapular nerve block (SSNB) with 5 mL bupivacaine 0.5%, then single shot US-guided costoclavicular block (CCB) with 10 ml bupivacaine 0.5%.
  Interventions: Procedure: Suprascapular Nerve Block with 5ml bupivicaine 0.5%; Procedure: costoclavicular Block 10ml bupivicaine 0.5%
- Interscalene brachial plexus block (Active Comparator): Single shot US-guided interscalene brachial plexus block (ISBPB) with 15 mL bupivacaine 0.5%.
  Interventions: Procedure: Interscalene Brachial Plexus Block 15ml bupivicaine 0.5%

INTERVENTIONS:
Procedure: Suprascapular Nerve Block with 5ml bupivicaine 0.5% — The patient lies supine with the head turned to the contralateral side to the block. Using a linear high-frequency ultrasound probe, the proximal suprascapular nerve is visualized before it turns toward the suprascapular notch. It is blocked using 5mL of bupivicaine 0.5%.
  Other Names: SSNB
  Arms: suprascapular nerve block with costoclavicular infraclavicular
Procedure: costoclavicular Block 10ml bupivicaine 0.5% — transverse ultrasound imaging of the medial infraclavicular fossa to identify the cords of the brachial plexus at the costoclavicular space (CCS) then inject 10ml bupivicaine 0.5%
  Other Names: CCB
  Arms: suprascapular nerve block with costoclavicular infraclavicular
Procedure: Interscalene Brachial Plexus Block 15ml bupivicaine 0.5% — The patient lies supine with the head turned to the contralateral side to the block. Using a linear high-frequency ultrasound probe, the interscalene groove is visualized along with the roots of the brachial plexus. The block is performed with 15mL of bupivacaine 0.5%.
  Other Names: ISBP
  Arms: Interscalene brachial plexus block

SUMMARY:
Postoperative analgesia for shoulder surgery is typically achieved by providing an interscalene brachial plexus block. However, a very common side effect of this block is hemi-diaphragmatic paralysis, a state which may not be tolerated in patients with pulmonary conditions such as COPD. Recently, clinicians have explored new ways to provide satisfactory analgesia while minimizing the pulmonary side effects of the interscalene nerve block. One of these solutions might be to offer the patient a suprascapular nerve block combined to a costoclavicular block. Since these blocks are performed lower in the neck or under the clavicle, the phrenic nerve is less likely to be blocked. Thus, fewer respiratory side effects have been reported when using such blocks. This prospective observational study will evaluate the patient response to surgical stimuli and the opioid requirements intraoperatively in patients undergoing shoulder arthroscopies with either a supraclavicular and costoclavicular blocks or an interscalene block.

Study Design: Prospective, randomized open label non-inferiority trial. Subject Population: Adults scheduled to undergo elective shoulder arthroscopy Sample Size: 50 patients Study Duration: Starts February 2020 - Ends February 2021 - Interim analysis at 30 patients Study Center: Assuit university hospital

DETAILED DESCRIPTION:
The main hypothesis of this study is that the suprascapular block combined with a costoclavicular block is not inferior to the interscalene brachial plexus block in terms of postoperative analgesia. Inverstigators postulate that postoperative pain score will not differ significantly in patients who receive either block.

secondary objectives will consist in looking at the differences in intraoperative anesthetic consumption, postoperative opioid consumption, arm motor block, diaphragmatic paresis, patient satisfaction and time for readiness to discharge from PACU. investigators hypothesize that these outcomes will be similar in both groups, with the exception of a potential reduction in arm motor block and diaphragmatic paresis in the combined suprascapular and costoclavicular block group.

After having obtained institutional ethics board approval of the study, patients older than 18 years old, scheduled for a first elective shoulder arthroscopy under general anesthesia will be screened in the pre-anesthesia clinic. patients will be approached and the whole study procedures will be explained extensively. Interested patients will be invited to sign the consent form .Patients will have the right to opt out at any time. The investigators will meet the patients again on the morning of the surgery to address any concerns. After consent, a study number will be allocated to the patient in ascending order.

Two groups will be evaluated:

* Group A: single shot US-guided suprascapular nerve block with 5 mL bupivacaine 0.5%, then single shot US-guided costoclavicular block with 10 ml bupivacaine 0.5%.
* Group B: single shot US-guided interscalene brachial plexus block with 15 mL bupivacaine 0.5%.

Tests will be done to evaluate the nerve block-induced loss of sensation to ice prior to entering the operating room (OR). Diaphragmatic excursion will be evaluated using an abdominal curvilinear ultrasound probe, and will be classified as being normal, paradoxical or immobile. Normal motion is caudad movement during inspiration. Paradoxical motion is cephalad movement during inspiration.

Once in the operating room, all routine monitors are connected.. Both study monitors are switched on and will record their respective indices continuously for the duration of the anesthesia. General anesthesia will be induced with propofol (1-2 mg/kg IV), fentanil (1 µg/kg IV bolus) and cis-atracium (0.1-0.2 mg/kg IV; ). A bolus of dexamethasone 4mg IV will be administered after induction of general anesthesia.

Patients will also have received oral acetaminophen 1g preoperatively. Intubation with an endotracheal tube is performed once the patient is adequately paralyzed . All drugs are given according to the adjusted body weight of the patient. This is calculated with Robinson's formula: where TBW is total body weight and IBW is ideal body weight (21-22). Immediately after intubation, anesthesia is maintained with isoflurane . At the end of anesthesia, Emergence and extubation are done in the OR. All times (start skin closure, start dressing, stop isoflurane) will be precisely reported in the CRF.

ELIGIBILITY:
Inclusion Criteria:

ASA status 1,2,3.

* Age 18 years or older
* Elective shoulder arthroscopic surgery under general anesthesia and nerve block performed preoperatively

Exclusion Criteria:

* Serious cardiac arrhythmias (including atrial fibrillation) or unstable coronary artery disease.
* Coagulation disorders.
* Patient refusal.
* Anatomical disorders and/or neuropathic disease.
* BMI above 40.
* History of substance abuse.
* Chronic use of psychotropic and/or opioid.
* History of psychiatric diseases needing treatment.
* Contraindications to nerve block for shoulder surgery.
* Allergy to fentanil or any drug in the study protocol.
* Failure of nerve block

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
pain scores on a scale from 0 to 10 | From entrance in PACU until PACU discharge e.g. up to 3 hours after surgery maximum
  PACU pain score from 1 to 10 which 1 indicate no pain and 10 maximum pain.
naluphine consumption postoperative | 2 hours postoperative
  use of naluphine for postoperative analgesia in mg by asking PACU nurse questionnaire

SECONDARY OUTCOMES:
Total dose fentanil in mcg | Intraoperative
  Total dose of fentanil in mcg from incision until wound dressing
Time to awakening in minutes | Intraoperative
  Time to awakening in minutes.
Time to extubation in minutes | Intraoperative
  Time to extubation in minutes.
Patient dyspnea on a scale from 0 to 10 in dyspnea scale | PACU e.g. up to 3 hours after surgery maximum
  Patient dyspnea prior to PACU discharge on a scale from 0 to 10.
24h pain scores on a scale from 0 to 10 at rest (NPS) | Postoperative at H24, 24 hours after surgery
  24h pain scores, H24
Duration of motor block in minutes strength | Postoperative for day 1 H24 24hours after surgery
  Duration of motor block in minutes, as measured by time to return of normal grip strength.
TIME OF 1ST RESCUE ANALGESIC | 24 hour postoperative
  time of 1st dose of naluphine use postoperative

CONTACTS AND LOCATIONS:
Overall Officials: mohamed talaat mohamed, MD, Principal Investigator — Assiut University
Locations (1):
- Assuit University Hospital, Asyut, Egypt